CLINICAL TRIAL: NCT02663245
Title: INTEGRA Study: Intervention in Type 2 Diabetes Mellitus Patients With Poor Glycemic Control on Primary Health Care.
Brief Title: INTEGRA Study: Primary Care Intervention in Type 2 Diabetes Patients With Poor Glycaemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Àngels Molló, MD, PhD, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: P14/129
Record Dates: First submitted 2015-12-04; First posted 2016-01-26 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention 1 (Experimental): Diabetes specific consultation + multicomponent intervention aimed at professionals and patients
  Interventions: Other: Intervention 1
- Intervention 2 (Experimental): Multicomponent intervention aimed at professionals and patients minus the diabetes specific consultation.
  Interventions: Other: Intervention 2
- Control group (No Intervention): No intervention. Data of the control groups will be retrieved from the SIDIAP.

INTERVENTIONS:
Other: Intervention 1 — * Diabetes specific consultation
  * Basic training in clinical guidelines
  * Platform of communication for professionals
  * Training update to review and evaluate actual cases where the coaching strategy has been applied 2-hours training programme to update and review the training of month 0.
  * 7-hour training programme in group coaching for primary care professionals with a theoretical and practical approach.
  * Intervention based on text messaging to patients to remind them of strategies that promote behaviour change in relation to diabetes.
  Arms: Intervention 1
Other: Intervention 2 — * 7-hour training programme in group coaching for primary care professionals with a theoretical and practical approach.
  * Training update to review and evaluate actual cases where the coaching strategy has been applied 2-hour training programme to update and review the training of month 0.
  * Basic training in clinical guidelines.
  * Platform of communication for professionals.
  * Intervention based on text messaging to patients to remind them of strategies that promote behaviour change in relation to diabetes.
  Arms: Intervention 2

SUMMARY:
The intensification of the management for the control of glycaemia and other risk factors in patients with type 2 diabetes (DM2) results in a reduction of diabetes-related complications.

The strategy to increase the competences of primary care professionals to improve health care has been mainly prompted by the current context of limited resources and restricted access to specialty care.

This study aims to evaluate the effectiveness and cost-effectiveness of an integral intervention carried out by primary care professionals with the following components:

1. detection of patients with poor diabetic control;
2. introduction of a specific consultation on diabetes followed by virtual and telephone specialist support;
3. introduction of other measures to overcome patients and professionals barriers to treatment.

The main objective of the study is to determine if glycaemic control as measured by the mean concentration of HbA1c of poorly controlled patients improves when these patients are evaluated and treated in primary care under the integral strategy proposed in this study. The INTEGRA project also includes Phase 1 (qualitative research study), which is aimed at identifying viable strategies to suppress barriers to treatment; these strategies have been included to the intervention study (phase 2).

Phase 2 is a controlled, quasi-experimental intervention that involves 9 primary care centres of 3 regions (Lleida, Girona, Barcelona). The participants are patients with DM2 with poor glycaemic control that meet all the inclusion criteria and sign the informed consent. The intervention study will have three arms: (1) Control Group; (2) Intervention Group 1 (diabetes specific consultation + additional measures originated in phase 1; and (3) Intervention Group 2 (additional measures originated in phase 1).

Phase 1 has been conducted during the last 6 months previous to the initiation of the proposed intervention study and consisted of a qualitative design (individualized interviews with randomly selected patients in each of the participating centers); this qualitative study has contributed to design the final intervention applied on phase 2, particularly, implementing additional measures as coaching sessions to health professionals of the participating centers and automated messaging to patients with reminder and motivational objectives.

Phase 2 consists of a recruitment period of 6 months, followed by a 12-month follow-up for each patient

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of Type 2 DM according to criteria of the World Health Organisation of one or more years of disease duration.
* Age from 30 to 80 years.
* HbA1C ≥ 9% (DCCT) according to the last blood test carried out during the 12 months prior to inclusion in the study
* No changes in the treatment that can influence the main variable during the 3 months prior inclusion in the study.
* Accepting to participate in the study and signing of the informed consent form.

Exclusion criteria:

* Patient refuses to participate and any other condition that prevents signing the informed consent form.
* Other types of diabetes: Type 1 DM, gestational diabetes and diabetes secondary to other diseases.
* Pharmacological treatments that interfere with carbohydrate metabolism, such as steroids.
* Life expectancy under 2 years.
* Current treatment for cancer other than basocellular or epidermoid skin cancer.
* Severe mental disease and dementia.
* Heart failure Class III or IV (NYHA).
* Renal transplant or current treatment with dialysis.
* Alcohol and drug abuse.
* Pregnancy or intention to get pregnant.
* Breastfeeding.
* Chronic treatment with steroids; treatment with steroids during the 2 months prior inclusion in the study.
* Pharmacological treatment for weight loss during the 2 months prior to inclusion in the - study.
* Treatment with immunosuppressants.
* Haemoglobinopathies and chronic anaemia.
* Body Mass Index > 45 mg/kg2 (1)
* Participation in clinical trials for medicines.
* Patients with conditions that prevent follow up and completion of protocol.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Glycaemic control measured by HbA1c | 12 months

SECONDARY OUTCOMES:
lipid profile control as measured by the mean concentration of LDL-cholesterol, non-HDL cholesterol and triglycerides | 12 months
measurement of systolic blood pressure and of diastolic blood pressure | 12 months
control of chronic complications associated with type 2 diabetes according to the protocol of the CIH | 12 months
direct health costs of type 2 diabetic patients | 12 months
evaluation of patient satisfaction using spanish version of diabetes treatment satisfaction questionnaire (DTSQ) | 12 months
control of risk factors, smoking and exercise: Patient Activation Measure questionnaire | 12 months
evaluation of therapeutic inertia: specific questionnaire created by Redgedaps | 12 months
evaluation of quality of life using spanish version of diabetes quality of life questionnaire (EsDQOL) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Àngels Molló, MD, Principal Investigator — Institut Català de la Salut; Dídac Mauricio, MD, PhD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Laura Montero, Tàrrega, LLeida, Spain

REFERENCES:
- [Derived] Mollo A, Vlacho B, Gratacos M, Mata-Cases M, Rubinat E, Berenguera Osso A, Cos FX, Franch-Nadal J, Khunti K, Mauricio D; INTEGRA research group. A multicomponent health care intervention is associated with improved glycaemic control in subjects with poorly controlled type 2 diabetes compared with routine care: The INTEGRA study. Diabetes Obes Metab. 2023 Dec;25(12):3549-3559. doi: 10.1111/dom.15250. Epub 2023 Aug 22. PMID 37608473
- [Derived] Mollo A, Berenguera A, Rubinat E, Vlacho B, Mata M, Franch J, Bolibar B, Mauricio D. INTEGRA study protocol: primary care intervention in type 2 diabetes patients with poor glycaemic control. BMC Fam Pract. 2019 Feb 7;20(1):25. doi: 10.1186/s12875-019-0916-9. PMID 30732583